CLINICAL TRIAL: NCT06431295
Title: Human Performance Evaluation of a Digital Visual Acuity Device: Visual Acuity-001
Brief Title: Evaluation of a Digital Visual Acuity Device vs. Standard Visual Acuity Measurements
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Antonio J. Forte, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 23-007148
Record Dates: First submitted 2024-05-22; First posted 2024-05-28 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Visual Acuity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Digital Visual Acuity Test (Experimental): Subjects for an ophthalmological examination that includes a visual acuity examination at Mayo Clinic in Florida have a digital visual acuity test conducted with the FaceScan device.
  Interventions: Device: FaceScan

INTERVENTIONS:
Device: FaceScan — Digital visual acuity device built for iOS ("iPhone") that conducts an assessment of visual acuity using a combination of integrated light detection and ranging (LiDAR) and voice processing.

SUMMARY:
The purpose of this research is to validate and determine the accuracy of the experimental device when measuring visual acuity versus our standard visual acuity measurements and to gather voice recordings of letters to help build a special system that recognizes spoken letters.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years) who come to Ophthalmology Clinic.
* Willing and able to provide consent.

Exclusion Criteria:

* Individuals < 18 years of age.
* Unable to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2027-10-01 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Number of times the experimental device when measuring visual acuity agreed with standard visual acuity measurements | Baseline
  Number of subjects to have agreement between the visual acuity digital device and the clinical assessment

SECONDARY OUTCOMES:
Voice samples | Baseline
  Total number of voice samples collected of spoken letters

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Forte, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No